CLINICAL TRIAL: NCT06162143
Title: Real World Evaluation of the Effect of Gelsectan® in Low Anterior Resection Syndrome Patients: a Pilot Prospective Case-series Pilot Study (GeLAR)
Brief Title: Effect of Gelsectan® in the Treatment of Low Anterior Resection Syndrome
Acronym: GeLAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 097-2022
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Low Anterior Resection Syndrome; Rectal cancer; xyloglucans; xylo-oligosaccharides
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gelsectan®: Patients in the Gelsectan® cohort will receive one capsule of Gelsectan® twice a day (after lunch and dinner) for 28 days.
  Interventions: Device: Gelsectan®

INTERVENTIONS:
Device: Gelsectan® — Gelsectan® is a CE-marked class II device containing xyloglucans, xylo-oligosaccharides, pea proteins, and tannins from grape seeds extract, already used in Irritable Bowel Syndrome (IBS).

SUMMARY:
Low Anterior Resection Syndrome (LARS) is an intestinal disorder affecting patients undergoing rectal resection for rectal cancer. A possible therapeutic option may be Gelsectan®, a class II device used in Irritable Bowel Syndrome (IBS). The aim of this study is to evaluate the efficacy of Gelsectan® in improving the symptoms of LARS.

DETAILED DESCRIPTION:
Low Anterior Resection Syndrome (LARS) affects almost 70% of patients after rectal resection for rectal cancer and is characterized by intestinal symptoms including urgency, fractioned defecation, and fecal incontinence. LARS is clinically diagnosed using the LARS score: a score higher than 21 indicates the presence of LARS and a score higher than 30 indicates severe LARS. The treatment opportunities for LARS are limited and failure rates are high. Gelsectan® is a class II device containing xyloglucans, xylo-oligosaccharides, pea proteins, and tannins from grape seeds extract, resulting effective in improving intestinal symptoms in patients with diarrheic Irritable Bowel Syndrome (IBS). Given the symptomatic similarities between LARS and IBS, Gelsectan® may represent a valid first line treatment for LARS patients.

The objective of this study is to provide preliminary data to determine whether the administration of Gelsectan® may ameliorate the symptoms of LARS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old.
* Patients who underwent low rectal resection for rectal cancer and who closed the ileostomy at least three months before the screening visit.
* Patients with a LARS score ≥21 and/or clinically relevant symptoms of urgency, increased stool frequency, or fecal incontinence.
* Patients indicated to treatment with Gelsectan® according to the clinical judgment.
* Oncological chemotherapy or radiotherapy completed at least four weeks before the screening visit.
* Presence of a functional, intact anastomosis.
* Female patients of childbearing potential must agree to use a reliable method of contraception.

Exclusion Criteria:

* Known hypersensitivity to the investigational medicinal product (IMP).
* Any condition that, in the opinion of the investigator, may interfere with the study procedures.
* Significant anastomotic complications (e.g., strictures, fistula), which may impair the treatment efficacy.
* Pregnant or breastfeeding women.
* Inability to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult rectal cancer patients who underwent low rectal resection and ileostomy closure.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Low Anterior Resection Syndrome (LARS) score | 28 days after treatment initiation
  The median Low Anterior Resection Syndrome (LARS) score before and after the treatment with Gelsectan®. The Low Anterior Resection Syndrome (LARS) score ranges from 0 to 42, where 0 represent no LARS symtpoms and 42 represent major LARS symtpoms.

SECONDARY OUTCOMES:
Air incontinence | 28 days after treatment initiation
  The grade of flatus incontinence as measured on Low Anterior Resection Syndrome (LARS) score. The air incontinence domain ranges from 0 (no symtpoms) to 7 (severe symtpoms).
Stool incontinence | 28 days after treatment initiation
  The grade of stool incontinence as measured on Low Anterior Resection Syndrome (LARS) score. The stool incontinence domain range from 0 (no symtpoms) to 3 (severe symptoms).
Stool frequency | 28 days after treatment initiation
  The grade of stool frequency as measured on Low Anterior Resection Syndrome (LARS) score. The stool frequency domain ranges from 0 (regular frequency) to 5 (irregular frequency).
Defecation fractioning | 28 days after treatment initiation
  The grade of defecation fractioning as measured on Low Anterior Resection Syndrome (LARS) score. The defecation fractioning domain ranges from 0 (no symptoms) to 11 (severe symptoms).
Defecation urgency | 28 days after treatment initiation
  The grade of defecation urgency as measured on Low Anterior Resection Syndrome (LARS) score. The defecation urgency domain ranges from 0 (no symptoms) to 16 (severe symptoms).
Memorial Sloan Kettering Cancer Center Bowel Function Instrument (MSKCC-BFI) score | 28 days after treatment initiation
  The median Memorial Sloan Kettering Cancer Center Bowel Function Instrument (MSKCC-BFI) score before and after the treatment with Gelsectan®. The Memorial Sloan Kettering Cancer Center Bowel Function Instrument (MSKCC-BFI) score ranges from 0 (normal defecatory condition) to 68 (severe defecatory symptoms).
Major Low Anterior Resection Syndrome (LARS) proportion | 28 days after treatment initiation
  The difference in the proportion of patients with a severe Low Anterior Resection Syndrome score before and after the treatment, as defined by a Low Anterior Resection Syndrome (LARS) score equal to or higher than 30.
Diarrhea | 28 days after treatment initiation
  The difference in the proportion of patients reporting diarrheic feces before and after the treatment as evaluated by the Bristol scale

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD,PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No